CLINICAL TRIAL: NCT05330520
Title: Prospective, Open-Label, Non-Comparative, Study to Assess the Long Term Safety and Efficacy of Butterfly Medical Prostatic Retraction Device in Benign Prostatic Hyperplasia (BPH) Patients Who Completed 12 Months of Follow-Up Post Implantation (Continuation Study for Study BM-011-IL)
Brief Title: Long Term Safety and Efficacy of Butterfly Medical Prostatic Retraction Device in Benign Prostatic Hyperplasia (BPH) Patients Who Completed 12 Months of Follow-Up Post Implantation (Continuation Study for Study BM-011-IL)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butterfly Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BM-011-LT
Record Dates: First submitted 2022-03-28; First posted 2022-04-15 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: BPH; BOO - Bladder Outflow Obstruction; Enlarged Prostate (BPH)
Keywords: LUTS; Urinary obstruction; Retrograde ejaculation
MeSH Terms: conditions — Prostatic Hyperplasia; Retrograde Ejaculation | interventions — Replantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients Who Completed 12 Months of Follow-Up Post Butterfly Implantation (Experimental): Continuation study for Study BM-011-IL
  Interventions: Procedure: Butterfly Medical Prostatic Retraction Device ("the Butterfly device") removal/replacement

INTERVENTIONS:
Procedure: Butterfly Medical Prostatic Retraction Device ("the Butterfly device") removal/replacement — when necessary, the device may be removed or replaced easily through the urethra due to its minimal surface and easy release from the mucosa covering it.

SUMMARY:
This study evaluates the long term safety and efficacy of use of the Butterfly Medical's prostatic retraction device in Benign Prostatic Hyperplasia (BPH) Patients. The study follows patients implanted with the Butterfly device for up to 5 year after implantation.

The evaluations include recording of safety events and BPH related symptoms by Uroflowmetry tests, residual urine and International Prostate Symptom Score (IPSS) questionnaires. The study also assesses the sexual quality of life after implantation of the Butterfly device.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a noncancerous enlargement of the prostate gland that may restrict the flow of urine from the bladder.

BPH is a proliferative process of the cellular elements of the prostate, also referred as enlarged prostate. Cellular accumulation and gland enlargement may be due to epithelial and stromal proliferation, impaired pre-programmed cell death (apoptosis), or both. More recently, the voiding dysfunction that ensues from prostate gland enlargement and bladder outlet obstruction (BOO) has been generically termed lower urinary tract symptoms (LUTS). These entities overlap; not all men with BPH have LUTS, and, likewise, not all men with LUTS have BPH. The same can be said for BOO.

An estimated 50% of men demonstrate histopathologic BPH by age 60 years. This number increases to 90% by age 85 years; thus, increasing gland size is considered a normal part of the aging process (2-5).

Approximately half of those diagnosed with histopathologic BPH demonstrate moderate-to-severe LUTS. Clinical manifestations of LUTS include urinary frequency, urgency, nocturia (getting up at night during sleep to urinate), decreased or intermittent force of stream, or a sensation of incomplete emptying. Complications occur less commonly but may include acute urinary retention, impaired bladder emptying, or the need for surgery.

The Butterfly Medical Prostatic Retraction Device is a retraction device, specially designed to be delivered into the prostatic urethra and indicated to dilate the prostatic urethra in BPH patients. This device was specially designed to reduce most of the known complications of used urethral stents.

The current clinical study is aimed to investigate the long term technical performance and clinical usage of Butterfly Medical Prostatic Retraction Device, through a 4 year follow up period, as a continuation of study BM-011-IL which assessed the above for a duration of 12 month post implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Completed 12 months follow up under study BM-011-IL. A subject that missed one or more visits during BM-011-IL will be included, as long as the subject has collected data at 12 months follow up visit.
2. Provide signed informed consent to the continuation study and be willing and able to perform follow up visits and activities as described in the study protocol.

Exclusion Criteria:

1. Patients which participated in the BM-011-IL study and did not complete 12 months follow up visit under study BM-011-IL due to any reason

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious adverse events (SAEs) and adverse events (AEs) related to the Butterfly Device. | 60 month post procedure
  Serious adverse events (SAEs) and adverse events (AEs) related to treatment with the Butterfly Device.
Change in IPSS change in post implantation patients. | 60 month post procedure
  Evaluate the change in IPSS during the FU at each timepoints in comparison to baseline before treatment.

SECONDARY OUTCOMES:
Incidence of device extraction and re-treatment | 60 month post procedure
  Rate and Time to device removal and re treatment
Rate of sexual dysfunction | 60 month post procedure
  Retrograde ejaculation rate in comparison to rate before treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Ziv Medical Center, Safed